CLINICAL TRIAL: NCT03766204
Title: Relationship Between Circulating CircRNAs and MicroRNAs and Severity of Experimental and Clinical ALI/ARDS
Brief Title: The Role of Circulating CircRNAs and MicroRNAs in Acute Lung Injury
Acronym: TRCCMALI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaofan Xia, President, Changhai Hospital
Other Study IDs: 20181204
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: circRNAs; microRNAs
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ARDS patients and healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARDS patients: 137 patients were enrolled consecutively over a two-year time period (2017-2018) and identified as ARDS prospectively according to the Berlin definitions of the European Society of Intensive Care Medicine and American Thoracic Society on ARDS. Exclusion criteria were an age of less than 18 years, pregnancy, chronic obstructive pulmonary disease according to medical history and failure to obtain informed consent.
- Healthy volunteers: Forty healthy volunteers recruited from the general population who had no significant medical history and no medications were categorized as control patients.

SUMMARY:
Efforts to identify circulating factors that predict severity of acute lung injury/acute respiratory distress syndrome（ALI/ARDS）patients is unrevealing. The primary purpose of this study is to verify circRNAs and microRNAs might be potential novel ALI/ARDS biomarkers and could play roles in pathogenesis of ALI/ARDS.

DETAILED DESCRIPTION:
Acute lung injury (ALI) or acute respiratory distress syndrome (ARDS) is a devastating cause of morbidity and mortality characterized by alveolar epithelial and endothelial injury. Despite recent advances in pathogenetic mechanisms and therapy strategies of ALI, efforts to identify circulating factors that predict severity of ALI/ARDS patients have been unrevealing.

Circular RNAs (circRNAs) are a novel class of endogenous non-coding RNA with a covalently continuous closed-loop structure. Compared with traditional linear RNAs, circRNAs are more stable and resistant to RNase R due to the absence of 5' caps and 3' tails, which show clear advantages in acting as novel molecular biomarkers for many diseases. In addition, many studies have reported that circRNAs can bind to microRNAs (miRNAs), acting as "miRNA sponges" which are named competitive endogenous RNAs (ceRNAs), and can regulate gene expression at the transcriptional or post-transcriptional level. Evidence indicates that circRNAs play important roles in cancers and other diseases such as tuberculosis and intervertebral disc degeneration. As no published research has studied the expression and role of circRNAs in the pathology and pathogenesis of ALI/ARDS, the investigators aimed to validate the aberrant expression of circRNAs in ALI/ARDS and explore the potential pathological mechanism in which circRNAs are involved.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ALI/ARDS
* Informed consent was obtained from either the subjects themselves or from designated surrogates before enrollment in the study.

Exclusion Criteria:

* Patients who have chronic lung disease before enrollment.
* Patients who have severe organ dysfunction, autoimmune diseases and tumor.
* Women who are pregnant or breast-feeding.
* Patients who, in the opinion of the Investigator, have any other medical condition which renders the patient unable to complete the study or which would interfere with optimal participation in the study or produce significant risk to the patient.
* Patients participating in or planning to enroll in another clinical trial during the time of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without ARDS were screened from Changhai Hospital. Patients were enrolled consecutively over a 2-year time period (2017-2018). All enrolled patients with ALI met the American-European Consensus Committee criteria.In addition, healthy individuals were recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Receiving Mechanical Ventilation | up to 28 days
Fraction of Inspired Oxygen (FiO2)/Partial Arterial Oxygen Pressure (PO2) | up to 28 days
Acute Physiology and Chronic Health Evaluation (APACHE) II Scores | up to 28 days
  APACHE II scores range from 0 to 71. A higher values represent a worse outcome
plasma circRNAs | Day 3
plasma microRNAs | Day 3

SECONDARY OUTCOMES:
Length of Stay in the ICU | 1 year
Length of Hospital Stay | 1 year
Days of Unassisted Ventilation | 1 year
Death | up to 28

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-fan Xia, MD;PHD, Study Director — Department of Burn Sugery, Changhai Hospital
Locations (1):
- Department of Burn and Trauma Sugery, Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No